CLINICAL TRIAL: NCT00019669
Title: Immunization of Patients With Metastatic Melanoma Using a Recombinant Fowlpox Virus Encoding a GP100 Peptide Preceded by an Endoplasmic Reticulum Insertion Signal Sequence
Brief Title: Vaccine Therapy With or Without Interleukin-2 in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066961; NCI-99-C-0044; NCI-T98-0088; NCT00001800 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2004-08

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin

INTERVENTIONS:
Biological: aldesleukin
Biological: fowlpox virus vaccine vector
Biological: gp100 antigen

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells. It is not yet known whether combining melanoma vaccine with interleukin-2 is more effective than vaccine therapy alone in treating metastatic melanoma.

PURPOSE: Phase II trial to compare the effectiveness of melanoma vaccine and interleukin-2 with that of melanoma vaccine alone in treating patients who have metastatic melanoma that has not responded to previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the clinical response in patients with metastatic melanoma treated with immunization with recombinant fowlpox vaccine administered either intravenously or intramuscularly, with or without interleukin-2 (IL-2).
* Compare the immune response in patients before and after treatment with these regimens.
* Compare the toxicity profile of these regimens in these patients.

OUTLINE: This is a partially randomized study. Patients are randomized to 1 of 3 treatment cohorts.

* Cohort 1: Patients receive recombinant fowlpox virus encoding gp100 peptide (fowlpox vaccine) IV once every 4 weeks for up to 4 doses. (Closed to accrual as of 6/21/02.)
* Cohort 2: Patients receive fowlpox vaccine intramuscularly (IM) once every 4 weeks for up to 4 doses. (Closed to accrual as of 6/21/04.)
* Cohort 3 (for patients in need of immediate interleukin-2 [IL-2] and those with disease progression after treatment in cohorts 1 or 2): Patients receive fowlpox vaccine either IV or IM* once every 4 weeks for 4 doses and IL-2 IV every 8 hours for a maximum of 12 doses beginning 24 hours after fowlpox vaccine.

NOTE: *The IM route of administration was selected as the preferred route of administration from cohorts 1 and 2

* Expanded cohort 2 (open to accrual 7/19/02): Patients receive fowlpox vaccine IM once every 4 weeks for up to 4 doses. Upon disease progression, patients receive fowlpox vaccine as above and IL-2 IV every 8 hours for a maximum of 12 doses beginning 24 hours after fowlpox vaccine. (Closed to accrual 12/4/03.) In all cohorts, 3-4 weeks after the last injection, patients achieving a complete remission may receive a maximum of an additional 2 courses of therapy. Patients with responding disease may receive repeat vaccinations for up to 8 courses. Patients with no response or progressive disease in cohorts not receiving IL-2 may be treated with fowlpox vaccine and IL-2 as in cohort 3. Patients who are randomized to receive IL-2 may not receive additional IL-2 therapy.

PROJECTED ACCRUAL: A maximum of 84 patients (24 in cohorts 1 and 2, 19-33 in cohort 3, and 27 in expanded cohort 2) will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven metastatic melanoma that has failed standard treatment
* Measurable disease
* HLA-A-201 positive

PATIENT CHARACTERISTICS:

Age:

* 16 and over

Performance status:

* ECOG 0-2

Life expectancy:

* More than 3 months

Hematopoietic:

* WBC ≥ 3,000/mm^3
* Platelet count ≥ 90,000/mm^3
* No coagulation disorders

Hepatic:

* Bilirubin ≤ 1.6 mg/dL (less than 3.0 mg/dL for patients with Gilbert's syndrome)
* AST/ALT < 2 times normal
* Hepatitis B surface antigen negative

Renal:

* Creatinine ≤ 2.0 mg/dL

Cardiovascular:

* No major cardiovascular disease
* No cardiac ischemia by a stress thallium test or other comparable test*
* No myocardial infarction*
* No cardiac arrhythmias* NOTE: *In order to be eligible to receive interleukin-2 (IL-2)

Pulmonary:

* No major respiratory disease
* No obstructive or restrictive pulmonary disease* NOTE: *In order to be eligible to receive IL-2

Immunologic:

* No autoimmune disease
* No known immunodeficiency disease
* No primary or secondary immunodeficiency
* No allergy to eggs
* No active systemic infections
* HIV negative

Other:

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other active major medical illness* NOTE: *In order to be eligible to receive IL-2

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior gp100 vaccination

Chemotherapy:

* Not specified

Endocrine therapy:

* No concurrent steroids

Radiotherapy:

* Not specified

Surgery:

* Prior surgery for the malignancy allowed

Other:

* At least 3 weeks since other prior therapy for the malignancy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-10; Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Rosenberg, MD, PhD, Study Chair — NCI - Surgery Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States

REFERENCES:
- [Background] Rosenberg SA, Yang JC, Schwartzentruber DJ, Hwu P, Topalian SL, Sherry RM, Restifo NP, Wunderlich JR, Seipp CA, Rogers-Freezer L, Morton KE, Mavroukakis SA, Gritz L, Panicali DL, White DE. Recombinant fowlpox viruses encoding the anchor-modified gp100 melanoma antigen can generate antitumor immune responses in patients with metastatic melanoma. Clin Cancer Res. 2003 Aug 1;9(8):2973-80. PMID 12912944